CLINICAL TRIAL: NCT03336905
Title: Implementation of a Program Based on Adapted Physical Activity and Recommendations for Second Cancers Prevention for Teenagers and Young Adults With Cancer
Brief Title: Implementation of a Program Based on Adapted Physical Activity and Recommendations for Second Cancers Prevention for TYACs
Acronym: PREVAPAJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREVAPAJA
Record Dates: First submitted 2017-10-30; First posted 2017-11-08 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms
Keywords: Adolescent and young adult
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity and Prevention (Experimental): * co-construction of supervised and non-supervised physical activity sessions with a physical activity trainer
  * balance sheet (at diagnosis and 4 monthes+/- 2 months later) : IPAQ, QLQC30, 6-min walk test, anthropometric evaluation
  * meetings and phone calls after the physical activity program to assess patient perception and satisfaction, and provide information and recommendations for cancer prevention
  Interventions: Other: Physical activity program and prevention after cancer

INTERVENTIONS:
Other: Physical activity program and prevention after cancer — Providing a supervised and non-supervised physical activity program for adolescent and Young adult with cancer and improve awareness on cancer prevention recommendations (second cancer risk, healthy lifestyles...)

SUMMARY:
About 700 new cases of cancer are recorded each year among TYAC aged 15 to 25 years old in Rhône-Alpes region (France); more than 200 are treated and supported within the TYAC Department of the Institute of Hematology and Oncology Pediatrics (Centre Léon Bérard-Civil Hospice of Lyon). These patients survive from their disease in 80% of cases; they have six times more likely to develop a risk of second primary cancer (SCP) than their peers. This risk of SCP is multifactorial and varies depending on the type of first cancer, treatment received and the prevalence of risk factors (smoking, overweight, sedentary lifestyle, environmental exposures...). This project aims to implement a clinical program based on adapted physical activity (APA) and cancer prevention recommendations for TYAC during the active treatment period (4-6 months). The methodology used series of assessments of APA sessions and information meetings dedicated to cancer prevention and SCP risk recommendations. It mobilizes regularly the health care team of TYAC Department, TYAC associations, sports structures and associations involved in cancer prevention at the regional level. Assessment of TYAC satisfaction regarding the project, benefits in terms of exercise practice, and knowledge improvement on cancer prevention recommendations, are assessed throughout the program.

ELIGIBILITY:
Inclusion Criteria:

* With neoplasms, histologically confirmed
* Whose ability to participate in the APA intervention has been certified by a medical certificate issued by physician, the referring physician or the physician investigator
* Covered by a medical insurance
* Written, signed informed consent

Exclusion Criteria:

* Cons-indication to physical activity practice, at discretion of the investigator

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Score of physical activity | 12 months
  International Physical Activity Questionnaire

SECONDARY OUTCOMES:
Score of quality of life | 4 months
  QLQC30
Score of fatigue | 4 months
  Visual analogic scale
Weight | 4 months
Waist circumference | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Perrine MAREC-BERARD, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carretier J, Boyle H, Duval S, Philip T, Laurence V, Stark DP, Berger C, Marec-Berard P, Fervers B. A Review of Health Behaviors in Childhood and Adolescent Cancer Survivors: Toward Prevention of Second Primary Cancer. J Adolesc Young Adult Oncol. 2016 Jun;5(2):78-90. doi: 10.1089/jayao.2015.0035. Epub 2015 Dec 1. PMID 26812458
- [Background] Duval S, Carretier J, Boyle H, Philip T, Berger C, Marec-Berard P, Fervers B. [Life style and occupational factors and prevention of second primary cancers after childhood and adolescent cancer: Current state of knowledge]. Bull Cancer. 2015 Jul-Aug;102(7-8):665-73. doi: 10.1016/j.bulcan.2015.03.017. Epub 2015 May 1. French. PMID 25936990